CLINICAL TRIAL: NCT05191485
Title: Shared Decision Making in Patients With Lung Cancer After Surgery：a Molecular Testing Decision Aid Evidence Based Development Study
Brief Title: Shared Decision Making in Patients With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Jiangyou People's Hospital (Unknown); Wu Jieping Medical Foundation (Other); Chongqing Medical University (Other); The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Xing Wei, Doctor, Sichuan Cancer Hospital and Research Institute
Other Study IDs: CN-SDM-Lung 1 Part I
Record Dates: First submitted 2022-01-01; First posted 2022-01-13 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Surgery; Lung Adenocarcinoma
Keywords: Shared-decision making; Decision aid
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Patients of decision making need assessment: We will conduct semi-structured interviews with target patients and patients' representatives to assess their decisional needs. Decisional needs including difficult decision type /timing, unreceptive decisional stage, decisional conflict (uncertainty), inadequate knowledge & unrealistic expectations, unclear values, inadequate support & resources, and Personal & clinical needs. All interviews will be conducted one-to-one or one-to-many (including families) and be audio-recorded for further analysis. Written informed consent will be obtained prior to each interview.
  Nonrandom purposive sampling will be used to select key respondents to conduct in depth interview. Snowball sampling, where potential participants are asked to identify others who may be willing to participate, as well as convenience sampling, will be utilized. For patients, aiming for diversity regarding age, sex, education level and annual household income. All participants should be Chinese-speaking.
  Interventions: Other: Qualitative interviews
- Other stakeholders of decision making need assessment: We will conduct semi-structured interviews with other stakeholders to assess their decisional needs. All interviews will be conducted one-to-one and be audio-recorded for further analysis. Written informed consent will be obtained prior to each interview.
  Nonrandom purposive sampling will be used to select key respondents to conduct in depth interview. Snowball sampling, where potential participants are asked to identify others who may be willing to participate, as well as convenience sampling, will be utilized. For other stakeholders (including thoracic surgeons, nurses, psychoanalyst, hospital administrators, molecular testing company staffs and insurance company staffs), region, seniority, position, and attitude toward both molecular testing and SDM are considered. All participants should be Chinese-speaking.
  Interventions: Other: Qualitative interviews
- Participants of cognitive debriefing/alpha tests: The purpose of Alpha test is to test the understandability of Decision Aid for Lung Cancer Molecular Testing version 1.0 (DA_LCMT 1.0). All debriefing interviews will be conducted one-on-one with structured probing questions. Participants will be encouraged to comment on DA_LCMT 1.0 and give recommendations to replace any unclear wording. At the start, the interviewer will explain the aim of the study and the procedures of the cognitive debriefing to participants. Then a paper-based DA_LCMT 1.0 will be given to participants, and sufficient time will be guaranteed to allow them to read DA_LCMT 1.0. The cognitive debriefing interview will start afterwards, and participants will answer questions probing questions asked by interviewers about DA_LCMT 1.0. Each cognitive debriefing interview will last for about 20 minutes. DA_LCMT 2.0 will be generated after the completion of the cognitive debriefing (Alpha test).
  Interventions: Other: Qualitative interviews
- Patients of Field testing /β tests: Then the investigators will conduct the field testing (Beta test) with patient and clinician facing the decision in real time. The purpose of Beta test is to test the usability of DA_LCMT 2.0 in "real-world setting". Clinician and patients will use the DA_LCMT 2.0 for real-time decision making. The conversation of decision progress will be audio-recorded. After the decision is made by patients, structured interview will be conducted and audio-recorded separately between clinician and patients. All the field testing interviews will conducted one-on-one and written informed consent will be obtained prior to each interview. Each field testing interview will last for about 20 minutes.
  Interventions: Other: Qualitative interviews
- Clinician of Field testing /β tests: Then the investigators will conduct the field testing (Beta test) with patient and clinician facing the decision in real time. The purpose of Beta test is to test the usability of DA_LCMT 2.0 in "real-world setting". Clinician and patients will use the DA_LCMT 2.0 for real-time decision making. The conversation of decision progress will be audio-recorded. After the decision is made by patients, structured interview will be conducted and audio-recorded separately between clinician and patients. All the field testing interviews will conducted one-on-one and written informed consent will be obtained prior to each interview. Each field testing interview will last for about 20 minutes.
  Interventions: Other: Qualitative interviews

INTERVENTIONS:
Other: Qualitative interviews — We will conduct semi-structured interviews with target patients, patients' representatives and other stakeholders to assess their decisional needs. The cognitive debriefing interview will start afterwards, and participants will answer probing questions asked by interviewers about DA_LCMT 1.0. Then the field testing interviews will conducted one-on-one structured interviews.

SUMMARY:
The objective of this study is to develop a Decision Aid for Lung Cancer Molecular Testing (DA_LCMT) and to facilitate shared-decision making in patients who were diagnosed with lung adenocarcinoma by intraoperative frozen pathology about whether to conduct the molecular testing.

DETAILED DESCRIPTION:
Under the guidance by Ottawa Decision Support Framework (ODSF), International Patient Decision Aid Standards (IPDAS) and FDA guidance for Identify what is important to patients, the investigators use semi-structured interviews qualitative research methods to generate the decision making needs items of lung cancer patients who were diagnosed with lung adenocarcinoma by intraoperative frozen section pathology and other stakeholders (including thoracic surgeons, nurses, hospital administrators, molecular testing company staffs and insurance company staffs). Then modified Delphi will be used to develop the Decision Aid for Lung Cancer Molecular Testing version 1.0 (DA_LCMT 1.0). One-to-one structured interviews qualitative research methods will be used in the Cognitive debriefing (alpha tests) and Field testing (β tests) to revise and improve the DA_LCMT from version 1.0 to finally version 3.0. Descriptive statistics will be used to summarize the baseline characteristics of patients and other stakeholders. Qualitative data will be analyzed by the three steps proposed by grounded theory.

ELIGIBILITY:
Inclusion criteria:

Patients of decision-making need assessment:

1) age ≥ 18 years; 2) patients with primary invasive adenocarcinoma of lung diagnosed by intraoperative frozen pathological section; 3) have or have not made a decision on lung cancer molecular testing (whether to perform molecular testing or not).

Other stakeholders of decision-making need assessment:

1) age ≥ 18 years; 2) relevant work experience ≥ 2 years; 3) for thoracic surgeons and personnel in molecular testing companies: have previous experience in communicating with patients about molecular testing related to lung cancer targeted therapy; 4) for nurses, hospital administrators, and personnel in insurance companies: have a certain understanding of the decision-making process.

Patients of Cognitive debriefing/Alpha tests:

1) age ≥ 18 years; 2) patients with primary invasive adenocarcinoma of lung diagnosed by intraoperative frozen pathological section; 3) have made a decision on whether to perform lung cancer molecular testing or not.

other stakeholders of Cognitive debriefing/Alpha tests:

1) age ≥ 18 years; 2) relevant work experience ≥ 2 years; 3) for thoracic surgeons and personnel in molecular testing companies: have previous experience in communicating with patients about molecular testing related to lung cancer targeted therapy; 4) for nurses, hospital administrators, and personnel in insurance companies: have a certain understanding of the decision-making process.

Patients of field testing /Beta tests:

1) age ≥ 18 years; 2) patients with primary invasive adenocarcinoma of lung diagnosed by intraoperative frozen pathological section; 3) have not decided whether to perform lung cancer molecular testing or not.

Clinician of field testing /Beta tests:

1) age ≥ 18 years; 2) relevant work experience ≥ 2 years; 3) previous experience in communicating with patients about molecular testing related to lung cancer targeted therapy; and 4) voluntarily participated in this study.

Exclusion criteria:

Inability to understand the research content.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-random purposive sampling will be used to select key respondents to participate in in-depth interviews. Snowball sampling, where potential participants are asked to identify others who may be willing to participate, as well as convenience sampling, will be utilized. For patients, we will aim for diversity regarding age, sex, education level, and annual household income. For other stakeholders (including thoracic surgeons, nurses, psychoanalysts, hospital administrators, molecular testing company staff, and insurance company staff), the representativeness in region, seniority, position, and attitude toward both molecular testing and SDM will be considered.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The DA_LCMT 3.0 | 3 days
  The DA_LCMT 3.0 is the final version in this study which must conform to the International Patient Decision Aid Standards (IPDAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Cancer Hospital & Institute, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei X, Liu Y, Yu H, Dai W, Yang D, Zhang K, Sun J, Xu W, Gong R, Yu Q, Pu Y, Wang Y, Liao J, Mu Y, Zhang Y, Feng W, Pan Q, Li Q, Shi Q. Protocol of an iterative qualitative study to develop a molecular testing decision aid for shared decision-making in patients with lung cancer after surgery. BMJ Open. 2022 Sep 19;12(9):e061367. doi: 10.1136/bmjopen-2022-061367. PMID 36123064